CLINICAL TRIAL: NCT03460418
Title: Treatment of Humerus Fractures by a Multiloc Nail, Through a Minimally Invasive Procedure.
Status: Completed | Type: Observational
Sponsor: Tamas Illes (Other)
Responsible Party: Sponsor-Investigator, Tamas Illes, Head of Clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Multiloc
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Humeral Fractures
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multiloc nail: Fracture treated with a Multiloc nail (patients treated between 2012 and 2017)
  Interventions: Other: Phone contact
- Philos plate: Fracture treated with a Philos plate (patients treated between 2012 and 2017)
  Interventions: Other: Phone contact
- arthroplasty: Fracture treated by arthroplasty (patients treated between 2012 and 2017)
  Interventions: Other: Phone contact

INTERVENTIONS:
Other: Phone contact — Assessment of the different outcomes by means of a phone contact

SUMMARY:
Proximal humerus fractures are more common in older people. They can be caused by a minor trauma on an osteoporotic bone.

Non- or little-displaced proximal humerus fractures are treated orthopedically. When the displacement is more important, the choice of the treatment is crucial and the algorithm of treatment is in permanent evolution. The technology and design of the implants and the operative techniques of osteosynthesis and arthroplasty have evolved. Patients live longer, they lead a more active life and their expectations have changed. The goals of the treatment should be an increase in shoulder function and a decrease in treatment failure.

This study analyzes the results of the treatment by intramedullary osteosynthesis using a Multiloc nail from Synthes between 2012 and June 2017. The study will compare the functional results obtained after fixation by a Multiloc nail, a Philos plate or arthroplasty.The functionality of the shoulder and the quality of life will be evaluated according to the type of treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients being treated for a proximal humerus fracture within the CHU Brugmann hospital between 2012 and 2017.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients beeing treated for a proximal humerus fracture within the CHU Brugmann hospital between 2012 and 2017.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Fracture classification (AO) | one year
  Fracture classification according to the "Müller AO Classification of fractures - long bones"
Fracture classification (NEER) | one year
  Fracture classification according to the "Neer classification of proximal humeral fractures"
Dash score | one year
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score is computed according to this formula: ([(sum of n responses)/n] -1)(25) where n represents the number of completed items. A higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability.The score ranges from 0 (no disability) to 100 (most severe disability).
Constant score | one year
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
QoL 36 | one year
  The QoL 36 quality of life questionnaire consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Victorien Gauchez, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No